CLINICAL TRIAL: NCT03894527
Title: Impact of Acute Exercise on Vascular Insulin Sensitivity in Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: American College of Sports Medicine (Other)
Responsible Party: Principal Investigator, Steven K. Malin, PhD, Assitant Professor, University of Virginia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 19060
Record Dates: First submitted 2019-03-05; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Acute Exercise; Endothelial Function; Simple Obesity; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Subjects with simple obesity will complete 2 different testing conditions in a counterbalanced order with at least one week between conditions.
  10-12 hrs post test condition the subject will report for a Euglycemic-Hyperinsulinemic clamp study, where Flow Mediated Dilation (FMD) and Contrast Enhanced Ultrasound (CEU) will be performed.
  Interventions: Behavioral: Single Bout of Exercise; Behavioral: Control Condition
- Metabolic Syndrome (Active Comparator): Subjects with metabolic syndrome will complete 2 different testing conditions in a counterbalanced order with at least one week between conditions.
  10-12 hrs post test condition the subject will report for a Euglycemic-Hyperinsulinemic clamp study, where Flow Mediated Dilation (FMD) and Contrast Enhanced Ultrasound (CEU) will be performed.
  Interventions: Behavioral: Single Bout of Exercise; Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Single Bout of Exercise — An exercise condition, which will be walking at a moderate intensity (~70% VO2peak). Time will vary based upon individual fitness levels to burn ~400kcals (estimated 0.5 - 1hr). Oxygen consumption will be measured during exercise via a metabolic cart to confirm energy expenditure. Participants will then rest following the exercise procedure for 20 minutes. Between 20 and 45 minutes following exercise, oxygen consumption will be measured to understand and capture excess post-exercise oxygen consumption (EPOC). Following this, participants will be provided with a standardize dinner and snack to consume in the AMP lab.
Behavioral: Control Condition — A control (no-exercise) condition. Participants will report to the AMP lab to rest for the same duration as the exercise bout and consume the standardized dinner and snack.

SUMMARY:
Obesity is an independent risk factor for type 2 diabetes and cardiovascular disease. The increased prevalence of obesity worldwide is a major concern among the scientific and medical communities. Insulin resistance is a common factor associated with obesity, metabolic syndrome, hypertension, and type 2 diabetes. Individuals affected by these conditions often experience endothelial dysfunction as well. Insulin resistance provides a key link between metabolic syndrome risk factors and vascular disease. Development of strategies aimed at preventing vascular dysfunction and future disease caused by metabolic disturbances is needed. Although the relationship between obesity and various diseases is well known, the acute effects of insulin on vascular function in obese individuals have yet to be fully determined. Additionally, the effects of acute exercise on insulin-stimulated endothelial function are unknown. Exercise may be an effective and potent treatment that protects against endothelial dysfunction, insulin resistance, and future cardiometabolic disease commonly present with obesity. However, less attention has been placed on vascular insulin sensitivity. The purpose of this study is to test the hypothesis that a single bout of exercise increases insulin-stimulated blood flow at the macro- and micro-vasculature level in obese individuals with metabolic syndrome to similar levels as healthy obese control. Our laboratory has available non-invasive methods to quantify vascular function and the gold-standard technique for assessing insulin sensitivity (euglycemic-hyperinsulinemic clamp). The investigators will assess vascular function (flow-mediated dilation, post-ischemic flow velocity and contrast-enhanced ultrasound) as well as arterial stiffness (augmentation index and pulse wave velocity) before and at the end of the clamp protocol performed the morning following a bout of exercise and a control (no-exercise) condition in 1) metabolic syndrome and 2) obese adults. If our hypothesis is sustained, it will suggest that a key role of the vasculature exists in regulating insulin following exercise and will provide insight into the link between the vasculature, obesity, metabolic syndrome and cardiovascular disease and may confer decreased risk for cardiometabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 40-70 years
* Never diagnosed with type 2 diabetes and/or cardiovascular disease
* Not currently engaged in > 60 min/wk of exercise
* Inclusion criteria specific to health obese vs. metabolic syndrome potential participants:

  * Healthy Obese: (BMI ≥ 30 kg/m2 but ≤ 45 kg/m2) and no other metabolic syndrome risk factors, excluding waist circumference.
  * Metabolic Syndrome: (BMI ≥ 30 kg/m2 but ≤ 45 kg/m2) and must meet at least 3 out of 5 National Cholesterol Education Adult Treatment Panel III Metabolic Syndrome Criteria:

Increased waist circumference (≥102 cm in men; ≥88 cm in women) Elevated triglycerides (≥150 mg/dl) or currently taking medication (Rx) Reduced HDL-cholesterol (<40mg/dl in men, <50 mg/dl in women) or currently taking medication (Rx) High blood pressure (≥130 mmHg systolic or ≥85mmHg diastolic) or currently taking medication (Rx) Elevated fasting glucose (≥100 mg/dl)

Subject may participate if on the following drugs:

* Diuretics, ace-inhibitors and ARBs for treatment of hypertension
* Statins

Exclusion Criteria:

* Morbidly obese patients (BMI >45 kg/m2) and overweight/lean patients (BMI <30 kg/m2).
* Subjects who have not been weight stable (>2kg weight change in past 3 months).
* Currently participating in a regular exercise training program ( >30 min. of physical activity per day, >2 days/week)
* Medication or food supplement that is known to affect insulin sensitivity or endothelial function (TZDs, sulfonylureas, biguanides, alpha-glucosidase inhibitors, phosphodiesterase inhibitors, beta-blockers, alpha-blockers, fibrates, glucocorticoids, fish oil, allopurinol)
* Subjects with abnormal estimated glomerular filtration rate (eGFR).
* Hypertriglyceridemic (>400 mg/dl) subjects.
* Hypertensive (>160/100 mmHg)
* Subjects taking vasoactive medications also known to affect heart rate and rhythm (i.e. Ca++ channel blockers, nitrates, alpha- or beta-blockers).
* Subjects with a history of significant metabolic, cardiac, congestive heart failure, cerebrovascular, hematological, pulmonary, gastrointestinal, liver, renal, or endocrine disease or cancer that in the investigator's opinion would interfere with or alter the outcome measures, or impact subject safety.
* Smoking presently or in the past 1 year.
* HbA1c ≥ 6.5
* Subjects currently taking Metformin or any active weight suppression medication (e.g. phentermine, orlistat, lorcaserin, naltrexone-bupropion in combination, liraglutide, benzphetamine, diethylpropion, phendimetrazine)
* Pregnant (as evidenced by positive pregnancy test) or breastfeeding
* Subjects with contraindications to participation in an exercise program
* Known hypersensitivity to perflutren (contained in Definity)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Effect of single bout of exercise on FMD | Baseline clamp study
  Flow Mediated Dilation (FMD) as a percentage
Effect of single bout of exercise on CEU | Baseline Clamp Study
  Contrast Enhanced Ultrasound (CEU) as a percentage
Comparison of insulin stimulated FMD response | Through study completion, up to about 4 weeks
  Flow mediated dilation as a percentage of fasting values
Comparison of insulin stimulated CEU response | Through study completion, up to about 4 weeks
  Contrast Enhanced Ultrasound (CEU) as a percentage of fasting values

SECONDARY OUTCOMES:
Systemic Arterial stiffness | Through study completion, up to about 4 weeks
  Augmentation Index as a percentage
Central Arterial Stiffness | Through study completion, up to about 4 weeks
  Pulse wave velocity in m/s
Metabolic Flexibility | Through study completion, up to about 4 weeks
  Respiratory gases in fasted and insulin-stimulated states in arbitrary units
Fasting glucose | Through study completion, up to about 4 weeks
  Comparison of glucose collected at baseline in mg/dl
Fasting insulin | Through study completion, up to about 4 weeks
  Comparison of insulin collected at baseline in uU/ml
Free Fatty Acids | Through study completion, up to about 4 weeks
  Comparison of free fatty acids collected at baseline in mEq/L
Adiponectin | Through study completion, up to about 4 weeks
  Comparison of inflammatory in ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Steve Malin, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore JX, Chaudhary N, Akinyemiju T. Metabolic Syndrome Prevalence by Race/Ethnicity and Sex in the United States, National Health and Nutrition Examination Survey, 1988-2012. Prev Chronic Dis. 2017 Mar 16;14:E24. doi: 10.5888/pcd14.160287. PMID 28301314
- [Background] Huang PL. A comprehensive definition for metabolic syndrome. Dis Model Mech. 2009 May-Jun;2(5-6):231-7. doi: 10.1242/dmm.001180. PMID 19407331
- [Background] Roberts CK, Hevener AL, Barnard RJ. Metabolic syndrome and insulin resistance: underlying causes and modification by exercise training. Compr Physiol. 2013 Jan;3(1):1-58. doi: 10.1002/cphy.c110062. PMID 23720280
- [Background] Barrett EJ, Liu Z. The endothelial cell: an "early responder" in the development of insulin resistance. Rev Endocr Metab Disord. 2013 Mar;14(1):21-7. doi: 10.1007/s11154-012-9232-6. PMID 23306779
- [Background] Goodpaster BH, Sparks LM. Metabolic Flexibility in Health and Disease. Cell Metab. 2017 May 2;25(5):1027-1036. doi: 10.1016/j.cmet.2017.04.015. PMID 28467922
- [Background] DeFronzo RA, Sherwin RS, Kraemer N. Effect of physical training on insulin action in obesity. Diabetes. 1987 Dec;36(12):1379-85. doi: 10.2337/diab.36.12.1379. PMID 3315786
- [Background] Morrish NJ, Wang SL, Stevens LK, Fuller JH, Keen H. Mortality and causes of death in the WHO Multinational Study of Vascular Disease in Diabetes. Diabetologia. 2001 Sep;44 Suppl 2:S14-21. doi: 10.1007/pl00002934. PMID 11587045
- [Background] Barrett EJ, Wang H, Upchurch CT, Liu Z. Insulin regulates its own delivery to skeletal muscle by feed-forward actions on the vasculature. Am J Physiol Endocrinol Metab. 2011 Aug;301(2):E252-63. doi: 10.1152/ajpendo.00186.2011. Epub 2011 May 24. PMID 21610226
- [Background] Barrett EJ, Eggleston EM, Inyard AC, Wang H, Li G, Chai W, Liu Z. The vascular actions of insulin control its delivery to muscle and regulate the rate-limiting step in skeletal muscle insulin action. Diabetologia. 2009 May;52(5):752-64. doi: 10.1007/s00125-009-1313-z. Epub 2009 Mar 13. PMID 19283361
- [Background] Inyard AC, Clerk LH, Vincent MA, Barrett EJ. Contraction stimulates nitric oxide independent microvascular recruitment and increases muscle insulin uptake. Diabetes. 2007 Sep;56(9):2194-200. doi: 10.2337/db07-0020. Epub 2007 Jun 11. PMID 17563063
- [Background] Muniyappa R, Yavuz S. Metabolic actions of angiotensin II and insulin: a microvascular endothelial balancing act. Mol Cell Endocrinol. 2013 Sep 25;378(1-2):59-69. doi: 10.1016/j.mce.2012.05.017. Epub 2012 Jun 7. PMID 22684034
- [Background] Zhao Y, Vanhoutte PM, Leung SW. Vascular nitric oxide: Beyond eNOS. J Pharmacol Sci. 2015 Oct;129(2):83-94. doi: 10.1016/j.jphs.2015.09.002. Epub 2015 Sep 28. PMID 26499181
- [Background] Jahn LA, Hartline L, Rao N, Logan B, Kim JJ, Aylor K, Gan LM, Westergren HU, Barrett EJ. Insulin Enhances Endothelial Function Throughout the Arterial Tree in Healthy But Not Metabolic Syndrome Subjects. J Clin Endocrinol Metab. 2016 Mar;101(3):1198-206. doi: 10.1210/jc.2015-3293. Epub 2016 Jan 12. PMID 26756115
- [Background] Reynolds LJ, Credeur DP, Manrique C, Padilla J, Fadel PJ, Thyfault JP. Obesity, type 2 diabetes, and impaired insulin-stimulated blood flow: role of skeletal muscle NO synthase and endothelin-1. J Appl Physiol (1985). 2017 Jan 1;122(1):38-47. doi: 10.1152/japplphysiol.00286.2016. Epub 2016 Oct 27. PMID 27789766
- [Background] Penedo FJ, Dahn JR. Exercise and well-being: a review of mental and physical health benefits associated with physical activity. Curr Opin Psychiatry. 2005 Mar;18(2):189-93. doi: 10.1097/00001504-200503000-00013. PMID 16639173
- [Background] Sjoberg KA, Frosig C, Kjobsted R, Sylow L, Kleinert M, Betik AC, Shaw CS, Kiens B, Wojtaszewski JFP, Rattigan S, Richter EA, McConell GK. Exercise Increases Human Skeletal Muscle Insulin Sensitivity via Coordinated Increases in Microvascular Perfusion and Molecular Signaling. Diabetes. 2017 Jun;66(6):1501-1510. doi: 10.2337/db16-1327. Epub 2017 Mar 14. PMID 28292969
- [Background] Malin SK, del Rincon JP, Huang H, Kirwan JP. Exercise-induced lowering of fetuin-A may increase hepatic insulin sensitivity. Med Sci Sports Exerc. 2014 Nov;46(11):2085-90. doi: 10.1249/MSS.0000000000000338. PMID 24637346
- [Background] Shojaee-Moradie F, Baynes KC, Pentecost C, Bell JD, Thomas EL, Jackson NC, Stolinski M, Whyte M, Lovell D, Bowes SB, Gibney J, Jones RH, Umpleby AM. Exercise training reduces fatty acid availability and improves the insulin sensitivity of glucose metabolism. Diabetologia. 2007 Feb;50(2):404-13. doi: 10.1007/s00125-006-0498-7. Epub 2006 Dec 6. PMID 17149589
- [Background] Hwang MH, Lee S. Insulin resistance: vascular function and exercise. Integr Med Res. 2016 Sep;5(3):198-203. doi: 10.1016/j.imr.2016.06.001. Epub 2016 Jun 9. PMID 28462118
- [Background] Dawson EA, Green DJ, Cable NT, Thijssen DH. Effects of acute exercise on flow-mediated dilatation in healthy humans. J Appl Physiol (1985). 2013 Dec;115(11):1589-98. doi: 10.1152/japplphysiol.00450.2013. Epub 2013 Sep 12. PMID 24030665
- [Background] Malin SK, Rynders CA, Weltman JY, Jackson Roberts L 2nd, Barrett EJ, Weltman A. Endothelial function following glucose ingestion in adults with prediabetes: Role of exercise intensity. Obesity (Silver Spring). 2016 Jul;24(7):1515-21. doi: 10.1002/oby.21522. Epub 2016 May 25. PMID 27221649
- [Background] Hallmark R, Patrie JT, Liu Z, Gaesser GA, Barrett EJ, Weltman A. The effect of exercise intensity on endothelial function in physically inactive lean and obese adults. PLoS One. 2014 Jan 20;9(1):e85450. doi: 10.1371/journal.pone.0085450. eCollection 2014. PMID 24465565
- [Background] Tjonna AE, Rognmo O, Bye A, Stolen TO, Wisloff U. Time course of endothelial adaptation after acute and chronic exercise in patients with metabolic syndrome. J Strength Cond Res. 2011 Sep;25(9):2552-8. doi: 10.1519/JSC.0b013e3181fb4809. PMID 21747296
- [Background] Will PM, Walter JD. Exercise testing: improving performance with a ramped Bruce protocol. Am Heart J. 1999 Dec;138(6 Pt 1):1033-7. doi: 10.1016/s0002-8703(99)70067-0. PMID 10577432
- [Background] Coggins M, Lindner J, Rattigan S, Jahn L, Fasy E, Kaul S, Barrett E. Physiologic hyperinsulinemia enhances human skeletal muscle perfusion by capillary recruitment. Diabetes. 2001 Dec;50(12):2682-90. doi: 10.2337/diabetes.50.12.2682. PMID 11723050
- [Background] Clerk LH, Vincent MA, Jahn LA, Liu Z, Lindner JR, Barrett EJ. Obesity blunts insulin-mediated microvascular recruitment in human forearm muscle. Diabetes. 2006 May;55(5):1436-42. doi: 10.2337/db05-1373. PMID 16644702
- [Background] Newsom SA, Everett AC, Hinko A, Horowitz JF. A single session of low-intensity exercise is sufficient to enhance insulin sensitivity into the next day in obese adults. Diabetes Care. 2013 Sep;36(9):2516-22. doi: 10.2337/dc12-2606. Epub 2013 Jun 11. PMID 23757424